CLINICAL TRIAL: NCT04731493
Title: Effect on the Quality of Life of a Therapeutic Education Program in Patients With Marfan Syndrome: an Observational, Prospective and Multicenter Study
Brief Title: Effect on the Quality of Life of a Therapeutic Education Program in Patients With Marfan Syndrome
Acronym: MYLIFE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0505
Record Dates: First submitted 2020-12-03; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Marfan Syndrome
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- therapeutic Education Program: individual and group sessions will be set up with educational workshops specialized by age group (child / adolescent / transition / adult / entourage / parents), socio-administrative workshops, etc.
  The objectives will be adapted to each age group and to each patient individually.
  Interventions: Other: Therapeutic Education Program

INTERVENTIONS:
Other: Therapeutic Education Program — * needs assessment
  * educational group workshop
  * specialized workshops by age group: child / adolescent / transition / adult / entourage / separated parents and in parallel
  * socio-administrative workshop
  * individual summary (accompanied or not by his entourage / family)
  * satisfaction questionnaire

SUMMARY:
This is a before-after, observational, prospective, multicenter cohort study. The study will consist of 2 phases: an initial observational phase of a minimum of 3 months before the Therapeutic Education Program (TEP) intervention, then a phase of evolution analysis of at least 3 months.

DETAILED DESCRIPTION:
During the first observational phase, the quality of life assessment will be carried out 3 months apart without intervention. The data obtained during this first phase will make it possible to characterize the functional impact in patients, to verify the reproducibility of our evaluations, and to evaluate the spontaneous evolution of the parameters over a period of 3 months.

During the second phase of evolution analysis, the quality of life will be assessed at 3 month intervals (M9, M12) after the therapeutic Education Program (M6). The comparison between the evolution during the two phases, before and after the TEP will allow us to assess the benefits of the TEP.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 7 and 25 years old with Marfan Syndrome or related according to Ghent criteria
* For minors, no oral opposition from the holders of parental authority and consent of the minor.
* For adults, no oral opposition collected
* Patient affiliated to a social security scheme or equivalent

Exclusion Criteria:

* Inability of the patient to understand the content of the TEP sessions or the questionnaire about quality of life (non-French speaking, severe intellectual disability)
* Patient who has already participated in a TEP session for his pathology.
* Protected adult: patient under legal guardianship or curator protection

Ages: 7 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patient with Marphan Syndrom
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
quality of life of children and young adults with Marfan | Base line
  Answer to the question of PedsQL
quality of life of children and young adults with Marfan syndrome after therapeutic education program (ETP), | 3 months
  Answer to the question of PedsQL
quality of life of children and young adults with Marfan syndrome after therapeutic education program (ETP), | 9 months
  Answer to the question of PedsQL
quality of life of children and young adults with Marfan syndrome after therapeutic education program (ETP), | 12 months
  Answer to the question of PedsQL

CONTACTS AND LOCATIONS:
Overall Officials: Yves DULAC, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No